CLINICAL TRIAL: NCT01818180
Title: Effect of URELL(Cranberry Vaccinium Macrocarpon)Consumption on the Prevalence of Recurrent Urinary Tract Infection and Asymptomatic Bacteriuria During Pregnancy.
Brief Title: Urell and Pregnancy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Double
Other Study IDs: 2009/19
Record Dates: First submitted 2013-03-19; First posted 2013-03-26 (Estimated); Last update posted 2013-03-26 (Estimated); Status verified 2013-03

CONDITIONS: Urinary Tract Infection (UTI)
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Urell (Experimental)
  Interventions: Dietary Supplement: URELL
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: URELL
  Arms: Urell
Other: Placebo
  Arms: Placebo

SUMMARY:
Evaluation of the effect of URELL consumption on the occurrence of recurrent urinary tract infection (Acute cystitis, pyelonephritis and asymptomatic bacteriuria).

ELIGIBILITY:
Inclusion Criteria:

- Pregnant woman in her 4th gestational month or more, having urinary tract infection.

Exclusion Criteria:

* Pregnant woman with organic or functional urinary tract malformations
* Diabetic patients
* HIV positive

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2010-05; Primary Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Recurrence of Urinary tract infections | From the 4th gestational month till the end of pregnancy (about the 40th gestational week)

CONTACTS AND LOCATIONS:
Overall Officials: Jean Marc AYOUBI, PU-PH, Study Chair — Hôpital FOCH 40, rue Worth 92150 Suresnes
Locations (1):
- Hôpital FOCH, Suresnes, France